CLINICAL TRIAL: NCT02016027
Title: Pharmacological Effect of Carica Folia Mother Tincture in Healthy Individual's Blood Parameter.
Brief Title: Pharmacological Effect of Carica Papaya Leaves Mother Tincture in Healthy Individuals Blood Parameter
Acronym: CF2013
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fr Muller Homoeopathic Medical College (Other)
Responsible Party: Principal Investigator, Dr Nimai Chandra Dhole, Principal Investigator, Fr Muller Homoeopathic Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: carica 2013; NCD
Record Dates: First submitted 2013-11-21; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carica folia Arm (Experimental)
  Interventions: Drug: Carica folia

INTERVENTIONS:
Drug: Carica folia

SUMMARY:
AIMS & OBJECTIVES To evaluate the effectiveness of administering of Carica folia mother tincture to healthy individual's Platelet count.

Sample Details:- Students, Doctors and non-teaching staffs of Father Muller Homoeopathic Medical College are taken up for the study. A minimum of 60 persons will be selected and will be divided into two groups, Control & Experiment by lottery method.

Voluntary participation in the study is expected. 30 persons in each group. One group will receive Carica folia mother tincture and other group will receive placebo.

Complete Blood count including platelet count will be measured for all 60 subjects before commencing the study.

The drug namely Carica Folia mother tincture will be procured from Father Muller Homoeopathic Pharmaceutical Division which compiles with the standards of Homoeopathic Pharmacopeia of India.

Daily dosage -30 drops of Carica Folia mother tincture in 30 ml of distilled water morning and night for 3days.

On 4th day complete blood count including platelet count will be estimated for all 60 subjects.

Research Methodology and Statistics:

Pre &Post with Control Design is done. Data from the sample is collected and is subjected to Paired 't' test and unpaired 't' test.

HYPOTHESIS:-

Null hypothesis:

No significant changes in complete blood count and platelet count before and after the intervention.

Alternate hypothesis:

There is significant variation in complete blood count and platelet count before and the intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* Age group- 18yrs to 25yrs
* both sexes
* free from any type of medicinal agent at least 15 days before commence the intervention.

Exclusion Criteria:

* person suffering from any illnesses
* age group below 18yrs and above 25yrs.
* person taking any medicinal agents, vitamins or any kinds of supplements will not be considered as subject.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Increase in platelet count | 3 days

SECONDARY OUTCOMES:
Increase in Red Blood Cell count | 3 days